CLINICAL TRIAL: NCT00939172
Title: An Open Label, Phase I, Single Group Assignment Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of TTP607 Administered in Cycles of Five Daily One to Four Hour Infusions to Patients With Advanced Refractory Solid Malignancies
Brief Title: TTP607 in Refractory Solid Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: vTv Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0219
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancers; Lymphoma
Keywords: Advanced Refractory Solid Malignancies; Solid tumor; Lymphoma; TTP607
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TTP607 (Experimental)
  Interventions: Drug: TTP607

INTERVENTIONS:
Drug: TTP607 — 3.3 mg/m^2 given by central venous catheter over 1-4 hours, each day for 5 days in a row, for a 15 day cycle.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of TTP607 that can be given to patients with a solid tumor or lymphoma. The safety of TTP607 will also be studied.

Researchers will also do pharmacokinetic (PK) testing of TTP607. PK testing measures the amount of a drug in the body at different time points.

DETAILED DESCRIPTION:
The Study Drug:

TTP607 is designed to work by blocking the action of certain enzymes (proteins) in the blood that are responsible for abnormal growth of cancer cells. This may cause the cancer cells to eventually die.

Dose Level Assignment:

If you are found to be eligible to take part in this study, you will be enrolled in a group of 3-6 participants. The dose you receive will be based on when you join this study (on how many participants have been enrolled before you, and on the safety data that is available at that time). The first group of participants will receive the lowest dose of TTP607. Each new group of participants will receive the next highest dose of the study drug, as long as no intolerable side effects occur. This process will continue until the highest tolerable dose of TTP607 is reached. Once the highest tolerable dose is found, 12 additional participants will be enrolled and treated at that dose, so that researchers can learn more about the effects of the study drug on the tumor. Both you and your study doctor will know what dose of the study drug you are receiving.

Study Drug Administration:

Starting on Day 1 of Cycle 1, you will receive TTP607 by central venous catheter (CVC or central venous line). There are several types of central venous catheters. Each type of catheter is a flexible, long, thin tube that is inserted through a vein, under a local anesthetic, through a small cut in your chest (near your heart). Some chemotherapy drugs are not suitable to be given into the veins in your hand or arm, so these drugs must be given into a larger vein. The CVC may also be used for drawing blood samples that are needed regularly. Using the CVC for these blood draws will lower the need for repeated blood draws from your arm. TTP607 will be given over 1-4 hours depending on the dose you receive, each day for 5 days in a row, followed by a 10-day "rest period" (no study drug). This 15 days is considered 1 cycle.

Study Visits:

On Day 1 (All Cycles):

You will have the below tests/procedures during your study visits:

* Your vital signs will be taken.
* You will have blood (about 1-2 tablespoons each time) drawn and urine collected for routine tests.
* You will be asked about any other medications that you may be taking and any side effects you may have experienced since your last visit.
* You will have an ECG.
* You will have a brief physical exam and routine eye exam.
* You will have a computed tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET) scan to check the size of the tumor.
* You will complete a questionnaire (1 question only) to rate your quality of life over the past week. It should take about 1 minute to complete.
* Women who are able to have children will have a urine pregnancy test.

On Days 2-5 (All Cycles):

The following tests/procedures will be performed before the start of the study drug infusion:

* You will be asked about any side effects that you may have had since your last visit.
* Your weight will be measured.

After the infusion, your vital signs will be measured.

On Days 2-5 (Cycle 1):

You will have an ECG performed, and blood (about 2-3 teaspoons each time) and urine will be collected for routine tests.

On Days 8, 10, and 12 (Cycle 1):

You will have the below tests/procedures during your study visits:

* You will complete the questionnaire to rate your quality of life over the past week.
* You will be asked about any medications you may have taken since your last visit and if you have had any side effects from them.
* You will have an ECG (Day 8 only).
* You will have blood (about 2-3 teaspoons each time) and urine collected for routine tests.
* You will have a brief physical exam and routine eye exam.
* Your weight will be measured (Days 8 and 12).
* Your vital signs will be measured.

On Days 3 and 5 (Cycles 2 and 3):

You will have an ECG.

On Days 2, 3, and 5 (Cycles 2 and 3):

You will have blood (about 2-3 teaspoons each time) drawn and urine collected for routine tests.

On Days 8-12 (Cycles 2, 3, and Further Cycles):

At least once at some time between Days 8 and 12, you will return to the clinic for the following tests/procedures:

* You will complete the questionnaire to rate your quality of life over the past week (on Day 12 of even-numbered cycles).
* You will be asked about any medications you may have taken since your last visit and if you have had any side effects from them.
* You will have an ECG (Cycles 2 and 3).
* You will have blood (about 2-3 teaspoons each time) and urine collected for routine tests.
* You will have a brief physical exam and routine eye exam.
* Your weight and vital signs will be measured.

On Day 5 (Cycle 4 and Further Cycles):

You will have blood (about 2-3 teaspoons each time) and urine collected for routine tests.

PK Testing:

You will have blood (about 2-3 teaspoons each time) and urine samples collected at different times for PK testing of TTP607.

Cycle 1:

Days 1 and 5:

Blood will be drawn immediately before the infusion, at 30 minutes during the infusion, at 60 minutes immediately after the infusion, and at 15 minutes, 30 minutes, 45 minutes, and at 1, 2, 3, 4, and 6 hours after the infusion.

On Day 1, urine will be collected immediately before the infusion and within 3 hours, between 3 and 7 hours, between 7 and 12 hours, and between 12 and 24 hours after the infusion. On Day 5, urine will be collected before the infusion and within 3 hours and between 3 and 7 hours after the infusion.

Days 2, 3, and 4:

Blood will be drawn immediately before the infusion and at 1 hour after the end of the infusion. Urine will be collected immediately before the infusion and within 2 hours after the end of the infusion.

Day 8:

Blood will be drawn at any convenient time, and urine will be collected when you first arrive in the clinic.

Cycles 2 and 3:

Days 1 and 5:

Blood will be drawn before the infusion and at 1 and 2 hours after the infusion, and urine will be collected before the infusion and within 2 hours after infusion.

Days 8-12:

Blood will be drawn at any convenient time, and urine will be collected when you first arrive in the clinic.

Cycle 4 and Further Cycles:

Day 5:

Blood will be drawn 1 hour after the infusion, and urine will be collected immediately before the infusion and within 2 hours after the infusion.

Length of Study:

You will continue on this study, as long as the study doctor thinks it is safe to continue, the cancer does not get worse, and if no intolerable side effects occur. If you continue on to further cycles, you will be on the same study drug schedule and will have the same tests/procedures for study visits, though they may be performed less often.

End-of-Study Visit:

Once you are off this study for any reason, you will have an end-of-study visit about 30 days after your last dose of the study drug. During this visit, you will have the following tests/procedures:

* You will have a complete physical exam, including measurement of your vital signs.
* Your blood (about 2 teaspoons) will be drawn and urine collected for routine tests.
* You will have an ECG.
* You will complete the questionnaire to rate your quality of life over the past week.
* Women who are able to have children will have a blood (about 1 teaspoon) pregnancy test.

This is an investigational study. TTP607 is not FDA approved or commercially available. At this time, it is being used for research purposes only. Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

Inclusion:

1. Patients with pathologically confirmed advanced malignancy that is metastatic or unresectable and which is refractory to standard therapy or for which there is no standard therapy.
2. Measurable disease at baseline.
3. At least four weeks since the last dose of prior chemotherapy, radiation therapy, or investigational agents, six weeks if the last regimen included BCNU or mitomycin C, six weeks if the agent was an antibody, four weeks if a chimeric antibody. For targeted therapies such as Gleevec®, Tarceva®, Nexavar®, Iressa®, or Sutent® at least five half-lives need to have elapsed since the last dose. Patients must be recovered from the adverse effects of prior therapy at the time of enrollment.
4. Age >/=18 years, male or female patients.
5. Women of child-bearing potential or men whose sexual partners are women of child-bearing potential must agree to use two methods of adequate contraception (i.e., hormonal and barrier method of birth control) prior to study entry, for the duration of the study, and for 30 days after the last dose of study medication.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
7. Patients must have normal organ and marrow function as defined: leukocytes >/= 3,000/mcL; absolute neutrophil count >/=1,500/mcL; platelets >/= 100,000/mcL; total bilirubin </= 2.0 mg/dL; AST(SGOT)/ALT(SGPT) </= 2.5 x upper limit of normal; and creatinine </= 2.0 mg/dL
8. Patients must have an existing patent and viable central venous catheter, or have such a line inserted within 28 days prior to initiation of study drug.
9. Patients must be able to understand and willing to sign a written informed consent document and have the capacity to follow study instructions.

Exclusion Criteria:

1. Uncontrolled concurrent illness, including but not limited to: ongoing or active infection, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, life-threatening cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements and/or obscure study results. Patients with a history of myocardial infarction in the last three months are also excluded from the trial.
2. Patients with known brain metastases that are symptomatic
3. Patients with leukemias or myelodysplastic syndrome (MDS).
4. Patients who have undergone bone marrow or stem cell transplantation within the last 5 years.
5. A requirement, as judged by the Principal Investigator, for primary prophylaxis with colony stimulating factors based on an expectation by the investigator of a risk of febrile neutropenia of 20% or greater or clinical factors that predispose the patient to increased complications from prolonged neutropenia as discussed in the latest American Society of Clinical Oncology (ASCO) recommendations for the use of white blood cell growth factor guidelines.
6. Nursing or pregnant women.
7. Documented HIV, HBV or HCV infection.
8. Patients with hypersensitivity to compounds of similar chemical or biologic composition to TTP607 or constituents of the intravenous (i.v.) formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03

PRIMARY OUTCOMES:
Maximum Tolerated Dose | End of each 15 day cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J. Wheler, MD, Study Chair — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org